CLINICAL TRIAL: NCT00235196
Title: A Study to Evaluate the Clinical Effectiveness of a Collagen-ORC Antimicrobial Matrix in Full-Thickness, Neuropathic Diabetic Foot Ulcers
Brief Title: Evaluation of the Clinical Effectiveness of a Collagen-ORC Antimicrobial Matrix in Full-Thickness, Neuropathic Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 400-04-001
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2006-10

CONDITIONS: Foot Ulcer
MeSH Terms: conditions — Foot Ulcer

INTERVENTIONS:
Device: Collagen ORC Antimicrobial Matrix (CAM)

SUMMARY:
This is a randomized (1:1), prospective, open label, multicenter, comparative study to be examine the effectiveness of Collagen-ORC Antimicrobial matrix, a new wound dressing, on diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Ambulatory (i.e. walking is the primary method of mobilization. Crutches, walker, walking frame or other ambulation aids are permitted).
* Diagnosed Type 2 diabetic (i.e. not juvenile onset).
* Have a DFU on the plantar surface of either foot.
* Have a DFU of >4 wks but <6 months duration.
* Willing and capable of cooperating to the extent and degree required by the study protocol

Exclusion Criteria:

* Be < 1cm2 or >10cm2 in area, by planimetry.
* Demonstrate overt signs of infection.
* Be located on the dorsal, lateral, or posterior heel area of the foot (Change 2, Amendment 1).
* Have visible exposed bone or tendon.
* Have an adjacent thermal injury or wound of an etiology other than diabetes.
* Be within 5 cm of any other wound, regardless of etiology.
* Have received enzymatic debriding agents in the past 7 days.
* Have received topical antibiotic therapy in the past 7 days.
* Be less than 1 cm2 or exceed 10cm2 in area by planimetry, after debridement.
* Have exposed bone or tendon, after debridement

The study subject MUST NOT:

* Have received previous treatment for the study ulcer by this Investigator.
* Have more than 3 full thickness ulcers, in total.
* Be pregnant or nursing an infant
* Have a concurrent illness or condition which may interfere with wound healing, such as carcinoma, vasculitis, immune system disorders or connective tissue disorder.
* Be a known alcohol or drug abuser.
* Have received systemic corticosteroids, immunosuppressive or chemotherapeutic agents in the past 30 days.
* Have received radiotherapy, which includes the lower extremity, at any time.
* Have a marked Charcot foot or claw foot deformity which would limit the ability of the subject to wear or be compliant with the wearing of the standardized off-loading device used in this study.
* Have received an investigational drug or device in the past 30 days.
* Have a known hypersensitivity to bovine collagen, oxidized regenerated cellulose (ORC) or silver.
* Be unwilling or unable to be fitted or compliant with the wearing of an ulcer off-loading device.
* Known to be non-compliant or unlikely to complete the study.
* Have ABPI < 0.7, OR, if ABPI >1.0 and toe pressure >0.6.
* Have serum Creatinine > 3 mg/dL25. have Hgb A1C>9%

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2004-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Clinical effectiveness of CAM in DFU by comparing the reduction in wound area between 2 treatment groups.

SECONDARY OUTCOMES:
Rate of wound closure
Ease of use and adverse events
Wound odor
Quality of life
Wound characteristics

CONTACTS AND LOCATIONS:
Overall Officials: James Hart, MD, Study Director — Ethicon, Inc.
Locations (3):
- United States (3):
  - Wound Care Center, Fort Lauderdale, Florida
  - Foot and Ankle Institute of South Florida, South Miami, Florida
  - Penn North Centers for Advanced Wound Care, Warren, Pennsylvania